CLINICAL TRIAL: NCT00833872
Title: LEO 22811 - A Phase I, Double-Blind, Placebo-controlled, Single and Multiple Oral Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Healthy Subjects
Brief Title: LEO 22811 - A Phase 1, Double-Blind, Placebo-controlled, Single and Multiple Oral Dose Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LEO 22811-S21
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2016-03

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 22811 solution (Experimental)
  Interventions: Drug: LEO 22811
- placebo solution (Placebo Comparator)
  Interventions: Drug: placebo solution

INTERVENTIONS:
Drug: LEO 22811 — First-in-man
  Arms: LEO 22811 solution
Drug: placebo solution
  Arms: placebo solution

SUMMARY:
The purpose of this first-in-man trial is to determine the safety and tolerability of ascending single and multiple doses of LEO 22811 in healthy male subjects as well as to determine the safety and tolerability of single oral doses of LEO 22811 in healthy female subjects. The trial will be performed in two parts. In Part 1, single doses of LEO 22811 will be administered to healthy male and female subjects. In Part 2, multiple doses of LEO 22811 will be administered to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria: (in summary)

* Subjects will be Caucasian males or females of non-child bearing potential between 18 and 65 years of age
* Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria: (in summary)

* Women of childbearing potential
* Subjects with an infectious illness within 3 days prior to dosing
* Subjects with a history of tuberculosis
* Subjects who have received any prescribed systemic or topical medication (including natural/herbal medicines) within 14 days of the first dose administration
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration
* In Part 2, subjects who have received or been exposed to Cloroquine products, endoxan, or any immunomodulating agent (e.g. azathioprin) within one month prior to the start of dosing
* Subjects who are participating in a clinical study
* Subjects with a significant history of drug allergy or with a known or suspected hypersensitivity to any of the components of LEO 22811 as determined by the Investigator
* Subjects who have any clinically significant allergic disease (excluding non-active hayfever) as determined by the Investigator
* Subjects who have a supine blood pressure and supine pulse rate at screening higher than 150/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/40 mmHg and 50 bpm, respectively
* Subjects who have PR interval >= 200 ms, QTc(b) interval >450 ms (males) or > 470 ms (females), or who exhibit U waves of atrio-ventricular blocks at screening, based on 12-lead ECGs
* Subjects who consume more than 28 units (males) or more than 21 units (females) of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse
* Subjects who smoke more than 5 cigarettes or the equivalent in tobacco per day
* Subjects with a significant cardiac history (e.g. heart failure, hypokalemia, long QT syndrome)
* Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator
* Subjects who, in the opinion of their General Practitioner (GP) or the Investigator, should not participate in the study, including subjects suspected for whatever reason of not being able to comply with the requirements of the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of ascending single and multiple oral doses of LEO 22811 in healthy male subjects. | 4 days
To determine the safety and tolerability of single oral doses of LEO 22811 in healthy female subjects. | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Lee, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No